CLINICAL TRIAL: NCT03028129
Title: Primary Prophylaxis for Prevention of TB in Prison's Populations
Brief Title: Prevention of Tuberculosis in Prisons
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim analysis showed efficacy less than 2.5%.
Sponsor: Federal University of Mato Grosso (Other)
Collaborators: Oswaldo Cruz Foundation (Other)
Responsible Party: Principal Investigator, Roberto D Oliveira, PhD Student, Federal University of Mato Grosso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: U1111-1189-0829
Record Dates: First submitted 2016-12-05; First posted 2017-01-23 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Tuberculosis, Pulmonary; Antibiotic Prophylaxis
Keywords: Tuberculosis; Primary prevention; Prisoners; Controlled Clinical Trial; Isoniazid
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Each subject received two oral supervised weekly doses of isoniazid 900 milligrams.
  Interventions: Drug: Isoniazid 900 milligrams
- Control (Placebo Comparator): Each subject received two oral supervised weekly doses of placebo (oral tablet, without the active ingredient, similar in size, weight, color, taste and odor).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Isoniazid 900 milligrams — Oral tablet, with the isoniazid 900mg, given two weekly. The administration will be supervised.
  Other Names: Antibiotic Treatment
  Arms: Treatment
Drug: Placebo — Oral tablet, without the active ingredient, similar in size, weight, color, taste and odor.
  Other Names: Placebo Treatment
  Arms: Control

SUMMARY:
The purpose of this study is to determine if the isoniazid is effective in the prevention of tuberculosis in a prison population, exposed to the high endemicity of the disease.

DETAILED DESCRIPTION:
Despite being a known disease of mankind over 9000 years, tuberculosis (TB) is still a major public health problem in developing countries, mainly due to so-called highly endemic sites, such as prisons.

It is Infectious disease, with airborne transmission, TB can present both the active or latent form. Despite the biological aspect of transmission, unhealthy environmental conditions (room without direct sunlight, poor ventilation and overcrowded) and individual factors (malnutrition, immunosuppression, use of alcohol and other drugs) have significant influence on transferability and infectivity.

With the discovery of drugs active against Mycobacterium tuberculosis, it was observed a reduction of disease incidence in the world. Despite this declining incidence, World Health Organization (WHO) classifies TB as a public health problem due to the emergence of multidrug strains or extensively resistant to treatment, added to the cases of latent TB reactivation, observed with the advent of HIV/AIDS.

Studies show a direct relationship between the incidence of TB and the prison environment. Nevertheless, the presence of prisons in one location increases the incidence of this disease, indicating that there is an exchange of disease between the prison and the community.

Currently, control of TB in the prison system is based on the tracking of individuals with active TB and / or latent and, in their respective treatment. For the identification of individuals with active disease, it is necessary the recognition of respiratory symptoms (cough mainly) and sputum smear microscopy and sputum culture, and chest X-ray. As the search of individuals with latent form, must be carried to the skin test with Purified Protein Derived (PPD).

Most of the units of the Brazilian's prison system these diagnostic methods are not available and hence the transport of individuals for their realization is necessary, generating an additional cost, in most cases, unfeasible process execution.

With the completion of this study, it seek to determine the effectiveness of primary prophylaxis in the prison population in order to gather new scientific evidence, to bring affordable methods for the control of TB in prisons.

Despite advances in diagnosis and treatment TB, this is the third leading cause of death from infectious diseases worldwide (Naghavi et al, 2015). In 2015, the WHO estimated incidence of 9.6 million new cases of TB in the world, with about 1.1 million deaths. For Brazil it was estimated incidence of 44 cases per 100,000 (WHO, 2015). The incidence of TB has declined about 2% per year, but this rate is not homogeneous in the global context.

Brazil occupies the 22nd place in the ranking of the WHO with an estimated annual rate of 83,310 cases of the disease (Zumla et al, 2015). In the past seven years, it is estimated that the incidence declined only 0.7% (per year). A key factor in this slow progress in TB control in Brazil, and other emerging countries is the existence of high-risk subpopulations, including slums and prisons, which act as reservoirs and amplifiers for the transmission of the disease (Basu; Stückler; Mckee 2011; Dowdy et al, 2012). A recent systematic review showed that the average incidence of TB in the prison population can be up to 23 times that recorded in the general population (Baussano et al, 2010).

With the fourth largest prison populations in the world, is observed in Brazil, the increased incidence of TB among prisoners in the last seven years. Although prisoners represent only 0.3% of the population, the increase in the prison population over this period resulted in almost doubling the proportion of all TB cases that occur among prisoners (4.1% in 2007, 8, 1% in 2013).

The arrests are in an ideal environment for the spread of TB, since they show individuals users of tobacco and alcohol in high doses, in addition to drug abuse in overcrowded cells with poor ventilation and with limited access to care health and diagnosis of TB. Currently, the Ministry of Health recommends active search for TB at the entrance to the prison and once a year by chest X-ray. Due to the cost and logistics, most prisons do not adhere to this recommendation. There is also a clear recommendation not to use the tuberculin skin test or perform the treatment for latent tuberculosis. If the procedures for active case detection and / or prophylactic treatment would impact the high transmission in prisons is a question that still remains open (Al-Darraji; Kamarulzamn; Altice, 2012).

The concentration of cases of TB in prisons can represent both an obstacle and an opportunity to control the disease, depending on the effectiveness of interventions in these environments.

Preliminary studies show high annual rate of TB infection (26%) among the prison population of 12 penitentiaries of Mato Grosso do Sul. Besides the large burden of disease in this population is significant dispersion of the TB prison to the community (Sacchi et al, 2015). Cross-sectional studies show high yield annual screening for TB, however, the effectiveness of this measure combined with other interventions remains unclear (Ferreira et al, 1996; Fournet et al, 2006; Lemos et al, 2014; Vieira et al, 2010; Sanches et al, 2013; Walnut; Abrahão; Galesi, 2012; Kuhleis et al, 2012; Estevan; Oliveira; Croda, 2013). Due to the combination of high force of infection in prisons and short prison term, primary prophylaxis may be an effective intervention. This new approach has never been evaluated in the context of prisons in low and middle income countries; to assess the impact of program strategies for TB screening and prophylaxis, longitudinal data will be essential. Given the infrastructure that was created for long-term prospective studies in Brazil, there is an excellent opportunity to close the critical knowledge gaps that have been barriers to effective implementation of TB control in high transmission prisons.

ELIGIBILITY:
Inclusion criteria:

* Age above 18 and under 45 at the time of inclusion;
* Sign the informed consent form.

Exclusion criteria:

* Be indigenous;
* Active TB or previous use of isoniazid;
* Score Alcohol Use Disorders Identification Test ≥15.
* Reactive serology for HIV, hepatitis B and C;
* Reactive result for quantiferon, considering as positive the result of Tube 1 and / or Tube22 above 0.2 IU / mL;
* Liver enzymes (Aspartate aminotransferase and Alanate aminotransferase) three times the upper limit;
* History or treatment for epilepsy;

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 467 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flora MF Moreira, Graduate, Study Chair — MsC Student; Andrea SS Carbone, MsC, Study Chair — PhD student; Flavia PC Sacchi, MsC, Study Chair — PhD student; Paulo CP Santos, Graduate, Study Chair — MsC Student; Rafaele CP Araújo, MsC, Study Chair — PhD student; Alessandra C Leite, MsC, Study Chair — PhD student; Cassia B Reis, PhD, Study Chair — Pos doc Student; Valeria C Rolla, PhD, Study Chair — Professor; Jason R Andrews, PhD, Study Chair — Professor
Locations (1):
- Roberto Oliveira, Dourados, Mato Grosso do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banerjee A, Dubnau E, Quemard A, Balasubramanian V, Um KS, Wilson T, Collins D, de Lisle G, Jacobs WR Jr. inhA, a gene encoding a target for isoniazid and ethionamide in Mycobacterium tuberculosis. Science. 1994 Jan 14;263(5144):227-30. doi: 10.1126/science.8284673.
- [Background] Barry CE 3rd, Boshoff HI, Dartois V, Dick T, Ehrt S, Flynn J, Schnappinger D, Wilkinson RJ, Young D. The spectrum of latent tuberculosis: rethinking the biology and intervention strategies. Nat Rev Microbiol. 2009 Dec;7(12):845-55. doi: 10.1038/nrmicro2236. Epub 2009 Oct 26. PMID 19855401
- [Background] Basu S, Stuckler D, McKee M. Addressing institutional amplifiers in the dynamics and control of tuberculosis epidemics. Am J Trop Med Hyg. 2011 Jan;84(1):30-7. doi: 10.4269/ajtmh.2011.10-0472. PMID 21212197
- [Background] Baussano I, Williams BG, Nunn P, Beggiato M, Fedeli U, Scano F. Tuberculosis incidence in prisons: a systematic review. PLoS Med. 2010 Dec 21;7(12):e1000381. doi: 10.1371/journal.pmed.1000381. PMID 21203587
- [Background] BERNSTEIN J, LOTT WA, STEINBERG BA, YALE HL. Chemotherapy of experimental tuberculosis. V. Isonicotinic acid hydrazide (nydrazid) and related compounds. Am Rev Tuberc. 1952 Apr;65(4):357-64. doi: 10.1164/art.1952.65.4.357. No abstract available. PMID 14903503
- [Background] Brites D, Gagneux S. Old and new selective pressures on Mycobacterium tuberculosis. Infect Genet Evol. 2012 Jun;12(4):678-85. doi: 10.1016/j.meegid.2011.08.010. Epub 2011 Aug 17. PMID 21867778
- [Background] Brosch R, Gordon SV, Marmiesse M, Brodin P, Buchrieser C, Eiglmeier K, Garnier T, Gutierrez C, Hewinson G, Kremer K, Parsons LM, Pym AS, Samper S, van Soolingen D, Cole ST. A new evolutionary scenario for the Mycobacterium tuberculosis complex. Proc Natl Acad Sci U S A. 2002 Mar 19;99(6):3684-9. doi: 10.1073/pnas.052548299. Epub 2002 Mar 12. PMID 11891304
- [Background] Carbone Ada S, Paiao DS, Sgarbi RV, Lemos EF, Cazanti RF, Ota MM, Junior AL, Bampi JV, Elias VP, Simionatto S, Motta-Castro AR, Pompilio MA, de Oliveira SM, Ko AI, Andrews JR, Croda J. Active and latent tuberculosis in Brazilian correctional facilities: a cross-sectional study. BMC Infect Dis. 2015 Jan 22;15:24. doi: 10.1186/s12879-015-0764-8. PMID 25608746
- [Background] Comas I, Coscolla M, Luo T, Borrell S, Holt KE, Kato-Maeda M, Parkhill J, Malla B, Berg S, Thwaites G, Yeboah-Manu D, Bothamley G, Mei J, Wei L, Bentley S, Harris SR, Niemann S, Diel R, Aseffa A, Gao Q, Young D, Gagneux S. Out-of-Africa migration and Neolithic coexpansion of Mycobacterium tuberculosis with modern humans. Nat Genet. 2013 Oct;45(10):1176-82. doi: 10.1038/ng.2744. Epub 2013 Sep 1. PMID 23995134
- [Background] Dowdy DW, Golub JE, Chaisson RE, Saraceni V. Heterogeneity in tuberculosis transmission and the role of geographic hotspots in propagating epidemics. Proc Natl Acad Sci U S A. 2012 Jun 12;109(24):9557-62. doi: 10.1073/pnas.1203517109. Epub 2012 May 29. PMID 22645356
- [Background] Estevan AO, Oliveira SM, Croda J. Active and latent tuberculosis in prisoners in the Central-West Region of Brazil. Rev Soc Bras Med Trop. 2013 Jul-Aug;46(4):515-8. doi: 10.1590/0037-8682-1441-2013. PMID 23904084
- [Background] Ferreira MM, Ferrazoli L, Palaci M, Salles PS, Medeiros LA, Novoa P, Kiefer CR, Schechtmann M, Kritski AL, Johnson WD, Riley LW, Ferreira Junior OC. Tuberculosis and HIV infection among female inmates in Sao Paulo, Brazil: a prospective cohort study. J Acquir Immune Defic Syndr Hum Retrovirol. 1996 Oct 1;13(2):177-83. doi: 10.1097/00042560-199610010-00009. PMID 8862283
- [Background] Fournet N, Sanchez A, Massari V, Penna L, Natal S, Biondi E, Larouze B. Development and evaluation of tuberculosis screening scores in Brazilian prisons. Public Health. 2006 Oct;120(10):976-83. doi: 10.1016/j.puhe.2006.06.004. Epub 2006 Sep 11. PMID 16965796
- [Background] FOX HH. The chemical approach to the control of tuberculosis. Science. 1952 Aug 8;116(3006):129-34. doi: 10.1126/science.116.3006.129. No abstract available. PMID 14950210
- [Background] Hanson ML, Comstock GW, Haley CE. Community isoniazid prophylaxis program in an underdeveloped area of Alaska. Public Health Rep (1896). 1967 Dec;82(12):1045-56. No abstract available. PMID 4966218
- [Background] Hershkovitz I, Donoghue HD, Minnikin DE, Besra GS, Lee OY, Gernaey AM, Galili E, Eshed V, Greenblatt CL, Lemma E, Bar-Gal GK, Spigelman M. Detection and molecular characterization of 9,000-year-old Mycobacterium tuberculosis from a Neolithic settlement in the Eastern Mediterranean. PLoS One. 2008;3(10):e3426. doi: 10.1371/journal.pone.0003426. Epub 2008 Oct 15. PMID 18923677
- [Background] Kuhleis D, Ribeiro AW, Costa ER, Cafrune PI, Schmid KB, Costa LL, Ribeiro MO, Zaha A, Rossetti ML. Tuberculosis in a southern Brazilian prison. Mem Inst Oswaldo Cruz. 2012 Nov;107(7):909-15. doi: 10.1590/s0074-02762012000700012. PMID 23147148
- [Background] Lemos EF, Alves AM, Oliveira Gde C, Rodrigues MP, Martins ND, Croda J. Health-service performance of TB treatment for indigenous and non-indigenous populations in Brazil: a cross-sectional study. BMC Health Serv Res. 2014 May 23;14:237. doi: 10.1186/1472-6963-14-237. PMID 24885134
- [Background] MacIntyre CR, Kendig N, Kummer L, Birago S, Graham NM. Impact of tuberculosis control measures and crowding on the incidence of tuberculous infection in Maryland prisons. Clin Infect Dis. 1997 Jun;24(6):1060-7. doi: 10.1086/513632. PMID 9195058
- [Background] Martinson NA, Barnes GL, Moulton LH, Msandiwa R, Hausler H, Ram M, McIntyre JA, Gray GE, Chaisson RE. New regimens to prevent tuberculosis in adults with HIV infection. N Engl J Med. 2011 Jul 7;365(1):11-20. doi: 10.1056/NEJMoa1005136. PMID 21732833
- [Background] GBD 2013 Mortality and Causes of Death Collaborators. Global, regional, and national age-sex specific all-cause and cause-specific mortality for 240 causes of death, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Jan 10;385(9963):117-71. doi: 10.1016/S0140-6736(14)61682-2. Epub 2014 Dec 18. PMID 25530442
- [Background] Nerlich AG, Haas CJ, Zink A, Szeimies U, Hagedorn HG. Molecular evidence for tuberculosis in an ancient Egyptian mummy. Lancet. 1997 Nov 8;350(9088):1404. doi: 10.1016/S0140-6736(05)65185-9. No abstract available. PMID 9365482
- [Background] Nguyen L, Pieters J. Mycobacterial subversion of chemotherapeutic reagents and host defense tactics: challenges in tuberculosis drug development. Annu Rev Pharmacol Toxicol. 2009;49:427-53. doi: 10.1146/annurev-pharmtox-061008-103123. PMID 19281311
- [Background] Nogueira PA, Abrahao RM, Galesi VM. Tuberculosis and latent tuberculosis in prison inmates. Rev Saude Publica. 2012 Feb;46(1):119-27. doi: 10.1590/s0034-89102011005000080. Epub 2011 Dec 13. PMID 22252791
- [Background] Sacchi FP, Praca RM, Tatara MB, Simonsen V, Ferrazoli L, Croda MG, Suffys PN, Ko AI, Andrews JR, Croda J. Prisons as reservoir for community transmission of tuberculosis, Brazil. Emerg Infect Dis. 2015 Mar;21(3):452-5. doi: 10.3201/eid2103.140896. PMID 25642998
- [Background] Salpeter SR. Fatal isoniazid-induced hepatitis. Its risk during chemoprophylaxis. West J Med. 1993 Nov;159(5):560-4. PMID 8279152
- [Background] Sanchez A, Massari V, Gerhardt G, Espinola AB, Siriwardana M, Camacho LA, Larouze B. X ray screening at entry and systematic screening for the control of tuberculosis in a highly endemic prison. BMC Public Health. 2013 Oct 20;13:983. doi: 10.1186/1471-2458-13-983. PMID 24139204
- [Background] Sharma SK, Sharma A, Kadhiravan T, Tharyan P. Rifamycins (rifampicin, rifabutin and rifapentine) compared to isoniazid for preventing tuberculosis in HIV-negative people at risk of active TB. Cochrane Database Syst Rev. 2013 Jul 5;2013(7):CD007545. doi: 10.1002/14651858.CD007545.pub2. PMID 23828580
- [Background] Smieja MJ, Marchetti CA, Cook DJ, Smaill FM. Isoniazid for preventing tuberculosis in non-HIV infected persons. Cochrane Database Syst Rev. 2000;1999(2):CD001363. doi: 10.1002/14651858.CD001363. PMID 10796642
- [Background] Sreevatsan S, Pan X, Stockbauer KE, Connell ND, Kreiswirth BN, Whittam TS, Musser JM. Restricted structural gene polymorphism in the Mycobacterium tuberculosis complex indicates evolutionarily recent global dissemination. Proc Natl Acad Sci U S A. 1997 Sep 2;94(18):9869-74. doi: 10.1073/pnas.94.18.9869. PMID 9275218
- [Background] Steingart KR, Ng V, Henry M, Hopewell PC, Ramsay A, Cunningham J, Urbanczik R, Perkins MD, Aziz MA, Pai M. Sputum processing methods to improve the sensitivity of smear microscopy for tuberculosis: a systematic review. Lancet Infect Dis. 2006 Oct;6(10):664-74. doi: 10.1016/S1473-3099(06)70602-8. PMID 17008175
- [Background] Sterling TR, Villarino ME, Borisov AS, Shang N, Gordin F, Bliven-Sizemore E, Hackman J, Hamilton CD, Menzies D, Kerrigan A, Weis SE, Weiner M, Wing D, Conde MB, Bozeman L, Horsburgh CR Jr, Chaisson RE; TB Trials Consortium PREVENT TB Study Team. Three months of rifapentine and isoniazid for latent tuberculosis infection. N Engl J Med. 2011 Dec 8;365(23):2155-66. doi: 10.1056/NEJMoa1104875. PMID 22150035
- [Background] Temple ME, Nahata MC. Rifapentine: its role in the treatment of tuberculosis. Ann Pharmacother. 1999 Nov;33(11):1203-10. doi: 10.1345/aph.18450. PMID 10573321
- [Background] THOREN M, HINSHAW HC. Therapy of pulmonary tuberculosis with isoniazid alone and in combination with streptomycin and with para-amino-salicylic acid. Stanford Med Bull. 1952 Nov;10(4):316-8. No abstract available. PMID 13015302
- [Background] Urrego J, Ko AI, da Silva Santos Carbone A, Paiao DS, Sgarbi RV, Yeckel CW, Andrews JR, Croda J. The Impact of Ventilation and Early Diagnosis on Tuberculosis Transmission in Brazilian Prisons. Am J Trop Med Hyg. 2015 Oct;93(4):739-46. doi: 10.4269/ajtmh.15-0166. Epub 2015 Jul 20. PMID 26195459
- [Background] Vieira AA, Ribeiro SA, de Siqueira AM, Galesi VM, dos Santos LA, Golub JE. Prevalence of patients with respiratory symptoms through active case finding and diagnosis of pulmonary tuberculosis among prisoners and related predictors in a jail in the city of Carapicuiba, Brazil. Rev Bras Epidemiol. 2010 Dec;13(4):641-50. doi: 10.1590/s1415-790x2010000400009. PMID 21180853
- [Background] Zumla A, George A, Sharma V, Herbert RH; Baroness Masham of Ilton; Oxley A, Oliver M. The WHO 2014 global tuberculosis report--further to go. Lancet Glob Health. 2015 Jan;3(1):e10-2. doi: 10.1016/S2214-109X(14)70361-4. No abstract available. PMID 25539957
- [Background] Al-Darraji HA, Kamarulzaman A, Altice FL. Isoniazid preventive therapy in correctional facilities: a systematic review. Int J Tuberc Lung Dis. 2012 Jul;16(7):871-9. doi: 10.5588/ijtld.11.0447. Epub 2012 Mar 7. PMID 22410101
- [Background] Barrera, L. The basics of clinical bacteriology Tuberculosis (2007): 93-112.
- [Background] Daniel TM. The history of tuberculosis. Respir Med. 2006 Nov;100(11):1862-70. doi: 10.1016/j.rmed.2006.08.006. Epub 2006 Sep 1. PMID 16949809
- [Background] Porter JD, McAdam KP. The re-emergence of tuberculosis. Annu Rev Public Health. 1994;15:303-23. doi: 10.1146/annurev.pu.15.050194.001511. PMID 8054087
- [Background] Nunn P, Williams B, Floyd K, Dye C, Elzinga G, Raviglione M. Tuberculosis control in the era of HIV. Nat Rev Immunol. 2005 Oct;5(10):819-26. doi: 10.1038/nri1704. PMID 16200083
- [Background] Schluger NW, Rom WN. The host immune response to tuberculosis. Am J Respir Crit Care Med. 1998 Mar;157(3 Pt 1):679-91. doi: 10.1164/ajrccm.157.3.9708002. No abstract available. PMID 9517576
- See also: World Prison Brief: Brazil. — http://www.prisonstudies.org/country/brazil
- See also: Power calculator for binary outcome superiority trial. — https://www.sealedenvelope.com/power/binary-superiority

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were interviewed for eligibility criteria (age, race, alcohol use, comorbidities) and laboratory tests (HIV, hepatitis B and C, liver enzymes, interferon gamma dosing for tuberculosis antigens and active tuberculosis).
Pre-assignment Details: Study was discontinued at ninth month after interim analysis and showed efficacy in intervention group less than 2.5%
Groups:
- Control: Each subject received two weekly supervised oral doses of placebo, without the active ingredient, similar in size, weight, color, taste and odor.
Period: Overall Study
Arm/Group | Treatment | Control
Started | 258 | 209
Completed | 132 | 122
Not Completed | 126 | 87
Not completed — Adverse Event | 13 | 2
Not completed — Lost to Follow-up | 50 | 38
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 62 | 45

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of isoniazid or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 258 | 209 | 467
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (6.7) | 29.0 (7.1) | 29.1 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 258 | 209 | 467
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 9 | 31
  White | 130 | 109 | 239
  More than one race | 105 | 90 | 195
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 258 | 209 | 467

OUTCOME MEASURES:

1. Primary Outcome: Quantiferon TB Gold Plus (QIAGEN®) Conversion at the Premature Exclusion Visit.
Description: Number of participants who had a Quantiferon TB Gold Plus (QIAGEN®) score greater than or equal to 0.35 international units per milliliter, at the time of the premature exclusion visit, on all participants in the group.
Time Frame: up to 6 months
Population: All participants who received at least one dose of isoniazid or placebo and who had blood sample collected to QFT examination at premature exclusion visit.
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 132 | 122
participants | 49 | 77

ADVERSE EVENTS:
Time Frame: 9 months
Description: On the intervention days, all participants were asked about the presence of any unusual signs and / or symptoms. Data were recorded in a log containing start and end date, event description, degree and intervention performed.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/258 | 0/209
Serious Adverse Events (participants affected / at risk) | 1/258 | 1/209
Other Adverse Events (participants affected / at risk) | 190/258 | 109/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=258) | Control (N=209)
Elevated SGOT (Hepatobiliary disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=258) | Control (N=209)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 24 (24)
Dizziness (Nervous system disorders) | 27 (27) | 8 (8)
Gastric pain (Gastrointestinal disorders) | 27 (27) | 15 (15)
Headache (Nervous system disorders) | 30 (30) | 15 (15)
Malaise (General disorders) | 29 (29) | 7 (7)
Nausea (Gastrointestinal disorders) | 20 (20) | 4 (4)
Somnolence (Psychiatric disorders) | 20 (20) | 9 (9)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 12 (12)
Flu syndrome (Infections and infestations) | 7 (7) | 15 (15)

LIMITATIONS AND CAVEATS:
Loss to follow-up Interruption of the study Arms presented differential group allocation Statistical power to detect the primary endpoint was 73%, lower than estimated in our sample size calculation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT03028129/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT03028129/ICF_001.pdf